CLINICAL TRIAL: NCT05726799
Title: Use of Cryoenergy to Faciltate Myectomy in Hypertrophic Obstructive Cardiomyopathy: Comparison With the Classical Approach
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: CRYO-MOR
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Septal Hypertrophy; Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cryoenergy
  Interventions: Procedure: Cryo myectomy
- Classic Myectomy
  Interventions: Procedure: Myectomy

INTERVENTIONS:
Procedure: Cryo myectomy — Extended septal myecotmy using cryo energy
  Groups: Cryoenergy
Procedure: Myectomy — Classic surgical myectomy
  Groups: Classic Myectomy

SUMMARY:
In some patients, septal hypertrophy extends more distally, from the subaortic portion of the septum to the midventricular portion. In these patients, classic transaortic surgical myectomy may not be effective in removing the midventricular obstruction, resulting in a suboptimal surgical outcome. These patients may present recurrence of symptoms and not have an improvement in the prognosis related to the treatment of hypertrophic cardiomyopathy, in some cases determining the need for reoperation. Since 2015, our Institute has used a surgical technique that allows us to improve transaortic exposure of the interventricular septum, using a probe with application of cryoenergy the hypertrophic portion of the septum is hooked and in this way the myectomy can be extended more distally, performing a more complete removal of the myocardium.

The aim of this study is to compare the results obtained with classical myectomy compared to myectomy performed with the aid of cryoenergy.

The primary endpoint is the comparison in terms of mortality between patients undergoing classical myectomy versus those undergoing cryoenergy-assisted myectomy.

Secondary endpoints are: extent of myectomy, persistence of residual left ventricular outflow tract obstruction, persistence of mitral regurgitation related to systolic anterior motion of the mitral leaflets, occurrence of ventricular defect, and need for PM implantation.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥ 18 years)
* meeting the clinical and echocardiographic criteria that made them candidates for isolated myectomy or in combination with other surgical procedures:
* LV outflow tract instantaneous peak gradient >50mmHg at rest or during stimulation
* interventricular septum >16mm,
* NYHA functional class III-IV, despite maximal medical therapy
* operated in San Raffaele Hospital with classic or cryo myectomy between 2015 and 2018.

Exclusion Criteria:

* extent of myectomy not reported in the operative report;
* left ventricular outflow tract gradient not reported in pre- or postoperative echocardiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing a myectomy due to obstructive hypertrophyc cardiomyopathy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No